CLINICAL TRIAL: NCT00300794
Title: Effects of Ketamine On Precipitated Opioid Withdrawal Under General Anaesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vilnius University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROT N1 V1_5
Record Dates: First submitted 2006-03-07; First posted 2006-03-09 (Estimated); Last update posted 2006-11-14 (Estimated); Status verified 2006-11

CONDITIONS: Opiate Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Ketamine

INTERVENTIONS:
Drug: Ketamine

SUMMARY:
The purpose of this study is to determine whether low-dose ketamine infusion is effective in suppressing the symptoms of opiate withdrawal during rapid opiate antagonist induction (RAI).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed opiate dependence according to ICD 10 and/or DSM 4;
* Duration of substance abuse more than 1 year
* No or minor co-morbidities;
* Grade I-II according to physical status classification system of American Society of Anesthesiologists.

Exclusion Criteria:

* Current history of long acting opiate or poly-substance abuse;
* Acute medical or surgical condition;
* Pregnancy;
* Breastfeeding.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60
Dates: Start 2003-02; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Juozas Ivaskevicius, Prof., Study Director — Vilnius University Clinic of Anaesthesiology and Intensive Care; Tomas Jovaisa, MD, Principal Investigator — Vilnius University Clinic of Anaesthesiology and Intensive Care
Locations (1):
- Vilnius University Emergency Hospital, Vilnius, Lithuania

REFERENCES:
- [Result] Ivaskevicius J, Jovaisa T, Laurinenas G, Vosylius S, Sipylaite J, Badaras R. [Safety and effectiveness of opiate antagonist detoxification under general anesthesia]. Medicina (Kaunas). 2005;41(12):1011-8. Lithuanian. PMID 16401957
- [Result] Jovaisa T, Laurinenas G, Vosylius S, Sipylaite J, Badaras R, Ivaskevicius J. Effects of ketamine on precipitated opiate withdrawal. Medicina (Kaunas). 2006;42(8):625-34. PMID 16963828